CLINICAL TRIAL: NCT04392531
Title: Open, Controlled, Randomized Clinical Trial to Evaluate the Efficacy and Safety of Cyclosporine Plus Standard Treatment vs Standard Treatment Only in Hospitalized Patients With COVID-19 Infection
Brief Title: Clinical Trial to Assess Efficacy of cYclosporine Plus Standard of Care in Hospitalized Patients With COVID19
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FJD-COVID19-20-01
Record Dates: First submitted 2020-05-03; First posted 2020-05-19 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: COVID19 Infection
MeSH Terms: conditions — COVID-19 | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (control) (Active Comparator): The control group will consist on the standard treatment that patients will receive according to hospital standard of care protocol.
  Interventions: Drug: Standard treatment
- Group B (experimental) (Experimental): The experimental group will consist on cyclosporine added to the standard treatment that patients will receive according to hospital standard of care protocol.
  Interventions: Drug: Cyclosporine

INTERVENTIONS:
Drug: Cyclosporine — In the experimental group, cyclosporine will be started according to patient weight, and then increased depending on patient tolerance (monitoring renal function and blood pressure)
  Arms: Group B (experimental)
Drug: Standard treatment — Standard of care according to hospital protocol
  Arms: Group A (control)

SUMMARY:
The study hypothesis is that cyclosporine, added to standard treatment of hospitalized patients with COVID19 infection may improve their prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Women and men over 18 years old
2. Clinical diagnosis of COVID19 infection (to be subsequently confirmed by PCR or specific IgM isotype Ac and with entry criteria according to the protocol of action (see Annex 2)
3. Acceptance and signing of the consent for the study after having received the appropriate information.

Exclusion criteria

1. Known allergy or hypersensitivity to any of the medications included in the treatment arms or to any of their components.
2. Contraindication for the use of any of the medications included (*)

   * CsA: IR EST 4.5 (FG <30 ml / min according to the Cockcroft-Gault formula)
   * Antimalarials (Chloroquine, hydroxychloroquine): Retinopathy, Myasthenia gravis.
   * Lopinavir / ritonavir: severe liver failure
   * Remdesivir, darunovir-ritonavir
   * Doxycycline, Azithromycin
3. Kidney failure (Stages 4 and 5: GFR <30 ml / min according to the cockcroft-Gault formula).
4. Decompensated liver disease (Child-Pugh stages B or C) or chronic infection with virus B
5. Pregnancy or lactation
6. Age over 75 years
7. Participants in another clinical trial with medication in the 28 days prior to the start of recruitment. Participation in observational studies is allowed.
8. Refusal to participate
9. Patient with a poor state of health or nutrition who, in the opinion of the researcher, has sufficient criteria of severity to interfere with the development of the study or its conclusions
10. At the investigator's discretion, the patient's inability to understand or comply with the study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Severity Category | 12 days
  efficacy of the association of CsA with standard treatment in reducing the severity of COVID19 infection in hospitalized patients.

SECONDARY OUTCOMES:
Mortality Rate | through study completion, an average of 6 weeks
  efficacy of CsA in combination with standard treatment in reducing mortality
Number of Days in hospital | through study completion, an average of 6 weeks
  efficacy of CsA in combination with standard treatment in reducing days in hospital
Number of days in ICU beds | through study completion, an average of 6 weeks
  efficacy of CsA in combination with standard treatment in reducing days in ICU beds
Fio2 Needs | through study completion, an average of 6 weeks
  efficacy of CsA in combination with standard treatment in reducing FiO2 needs.
Adverse events rate | through study completion, an average of 6 weeks
  safety and tolerability of cyclosporine vs standard treatment administration
Change in CRP | every 48 hours from randomization until patient discharge, and at the end of study visit (14 days after discharge or 14 days after end of study treatment, depending of what applies)
  change from baseline in C reactive protein levels
Change in ferritin | every 48 hours from randomization until patient discharge, and at the end of study visit (14 days after discharge or 14 days after end of study treatment, depending of what applies)
  change from baseline in ferritin levels
Change in LDH | every 48h during hospitalization and end of study visit (14 days after discharge or 14 days after end of study treatment)
  change from baseline in LDH levels
Change in CPK | every 48 hours from randomization until patient discharge, and at the end of study visit (14 days after discharge or 14 days after end of study treatment, depending of what applies)
  change from baseline in Creatin phosphokinase levels
Change in D Dimer | every 48 hours from randomization until patient discharge, and at the end of study visit (14 days after discharge or 14 days after end of study treatment, depending of what applies)
  change from baseline in D Dimer levels
Change in IL-6 | Days 1, 8, 15 and end of study visit (14 days after discharge or 14 days after end of study treatment)
  change from baseline in IL-6 levels
Change in KL-6 | Days 1, 8, 15 and end of study visit (14 days after discharge or 14 days after end of study treatment)
  change from baseline in KL-6 levels
Change in Viral Load | Days 1,8,15 and end of study visit (14 days after discharge or 14 days after end of study treatment)
  COVID19 Viral load determination
Change specific antibodies | Days 1,8,15 and end of study visit (14 days after discharge or 14 days after end of study treatment)
  Specific IgG and IgM determination

CONTACTS AND LOCATIONS:
Overall Officials: Olga Sanchez Pernaute, MD, PhD, Principal Investigator — FUNDACION JIMENEZ DIAZ
Locations (7):
- Spain (7):
  - Complejo Hospitalario Universitario La Coruña, A Coruña, Galicia
  - Hospital Quiron La Coruña, A Coruña, Galicia
  - Hospital Rey Juan Carlos, Móstoles, Madrid
  - Hospital Infanta Elena, Valdemoro, Madrid
  - Hospital General de Villalba, Villalba, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Clinica Universitaria de Navarra, Madrid